CLINICAL TRIAL: NCT00479258
Title: Safety And Efficacy Of Exubera® (Inhaled Insulin) Compared With Subcutaneous Human Insulin Therapy In Children And Adolescents Ages 6-17 Years With Type 1 Diabetes Mellitus: A 12 Month, Outpatient, Randomized, Open Label, Parallel Group Comparative Trial.
Brief Title: Safety And Efficacy Of Exubera Compared With Subcutaneous Human Insulin Therapy In Children And Adolescents
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A2171083
Record Dates: First submitted 2007-05-24; First posted 2007-05-28 (Estimated); Results first posted 2008-11-03 (Estimated); Last update posted 2018-10-01 (Actual); Status verified 2018-08

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Exubera

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Inhaled insulin (Exubera) (Experimental)
  Interventions: Drug: Inhaled insulin (Exubera)
- Subcutaneous Insulin (subject's prescribed) (Active Comparator)
  Interventions: Drug: Subcutaneous Insulin (subject's prescribed)

INTERVENTIONS:
Drug: Inhaled insulin (Exubera) — Inhaled insulin with dose adjusted according to premeal blood glucose
  Arms: Inhaled insulin (Exubera)
Drug: Subcutaneous Insulin (subject's prescribed) — Subcutaneous insulin with dose adjusted according to premeal blood glucose
  Arms: Subcutaneous Insulin (subject's prescribed)

SUMMARY:
To assess the safety and efficacy of Exubera on pulmonary function and glycemic control in subjects ages 6-17 over a 1 year period.

DETAILED DESCRIPTION:
Pfizer announced in October 2007 that it would stop marketing Exubera. At that time recruitment for the pediatric study, A2171083, was placed on hold. Two subjects completed the informed consent/assent process and entered the A2171083 study but none received treatment. The first subject withdrew consent during the Baseline Run-in period which was prior to Randomization. The second subject screen failed at Visit 1. After this time, Nektar, the company from which Pfizer licensed Exubera, announced on April 9, 2008 that it had stopped its search for a new marketing partner. Accordingly, there will be no commercial availability of Exubera. As a result, study A2171083 was terminated and no further recruitment took place.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with Type 1 diabetes mellitus for more than 6 months.
* Males and females ages 6 to 17 years.
* Subjects should be receiving, or be able to tolerate, at a minimum a 3 unit pre prandial dose of short acting subcutaneous insulin.

Exclusion Criteria:

* Subjects using an insulin pump
* Smoking

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2007-10; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Buffalo, New York, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A2171083&StudyName=Safety%20And%20Efficacy%20Of%20Exubera%20Compared%20With%20Subcutaneous%20Human%20Insulin%20Therapy%20In%20Children%20And%20Adolescents

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Two subjects completed the informed consent/assent process and entered the A2171083 study but none received treatment. The first subject withdrew consent during the Baseline Run-in period which was prior to Randomization. The second subject screen failed at Visit 1. Location = UNITED STATES.
Pre-assignment Details: Pfizer announced in Oct 2007 that it would stop marketing Exubera. At that time recruitment was placed on hold. Nektar, the company from which Pfizer licensed Exubera, announced on April 9, 2008 that it had stopped its search for a new marketing partner. As a result, study A2171083 was terminated and no further recruitment took place.
Groups:
- Inhaled Insulin (Exubera); Subcutaneous Insulin (Subject's Prescribed): No subjects received study medication.
Period: Overall Study
Arm/Group | Inhaled Insulin (Exubera) | Subcutaneous Insulin (Subject's Prescribed)
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Inhaled Insulin (Exubera) | Subcutaneous Insulin (Subject's Prescribed) | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Customized [unit: subjects] — <18 years
Sex: Female, Male

OUTCOME MEASURES:

1. Primary Outcome: To Assess Pulmonary Safety and Glycemic Control of Exubera Over a 12 Month Controlled Period
Description: No subjects were dosed therefore no data collected.
Time Frame: 12 months
Population: No subjects were dosed therefore no participants for analysis.
Arm/Group | Inhaled Insulin (Exubera) | Subcutaneous Insulin (Subject's Prescribed)
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change From Baseline in Other PFT Parameters
Time Frame: 12 months
Reporting Status: Not Posted

3. Secondary Outcome: Slope From Baseline to Week 52 and Slope From Week 12 to Week 52 for FEV1 and FVC as a Percent of Predicted;
Time Frame: 12 months
Reporting Status: Not Posted

4. Secondary Outcome: Treatment Preferences.
Time Frame: 12 months
Reporting Status: Not Posted

5. Secondary Outcome: Change From Baseline in FVC
Time Frame: 12 months
Reporting Status: Not Posted

6. Secondary Outcome: Slope for Other PFT Parameters;
Time Frame: 12 months
Reporting Status: Not Posted

7. Secondary Outcome: Proportion of Subjects Achieving ADA Age Appropriate Guidelines for HbA1c
Time Frame: 12 months
Reporting Status: Not Posted

8. Secondary Outcome: Change From Baseline in Insulin Antibodies (microU/mL);
Time Frame: 12 months
Reporting Status: Not Posted

9. Secondary Outcome: Change From Baseline in Body Weight (kg), Height (cm), and Body Mass Index (BMI; kg/m2) and z Score (%);Dose of Insulin;
Time Frame: 12 months
Reporting Status: Not Posted

10. Secondary Outcome: Hypoglycemic Event Rates;
Time Frame: 12 months
Reporting Status: Not Posted

11. Secondary Outcome: 7 Point Home Glucose
Time Frame: 12 months
Reporting Status: Not Posted

LIMITATIONS AND CAVEATS:
Pfizer announced Oct07 it would stop marketing Exubera; recruitment placed on hold. Nektar, from which Pfizer licensed Exubera, announced April 9, 2008 it had stopped its search for a new marketing partner. Study terminated; no further recruitment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of <60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), <12 mo from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential info other than study results.